CLINICAL TRIAL: NCT00027833
Title: Pilot Phase II Study of Safety and Immunogenicity of an ALVAC-CEA/B7.1 Vaccine Administered With Chemotherapy, Alone or in Combination With Tetanus Toxoid, as Compared to Chemotherapy Alone, in Patients With Metastatic Colorectal Adenocarcinoma
Brief Title: Vaccine Therapy and Chemotherapy With or Without Tetanus Toxoid Compared With Chemotherapy Alone in Treating Patients With Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000069082; CPMC-14534; CPMC-BB-IND-9911; FCCC-01015; APL-COL13; NCI-G01-2033
Record Dates: First submitted 2001-12-07; First posted 2003-01-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2003-09

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Tetanus Toxoid; Fluorouracil; Irinotecan; Leucovorin

INTERVENTIONS:
Biological: ALVAC-CEA-B7.1 vaccine
Biological: tetanus toxoid
Drug: FOLFIRI regimen
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Tetanus toxoid may make tumor cells more sensitive to chemotherapy and vaccine therapy.

PURPOSE: Randomized phase II trial to study the effectiveness of chemotherapy and vaccine therapy with or without tetanus toxoid compared with chemotherapy alone in treating patients who have metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of ALVAC-CEA-B7.1 vaccine and chemotherapy, with or without tetanus toxoid, vs chemotherapy alone in patients with metastatic colorectal adenocarcinoma.
* Determine whether tetanus toxoid enhances the immune response in patients treated with the vaccine and chemotherapy.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive a priming dose of tetanus toxoid. Beginning 2 weeks later, patients receive tetanus toxoid and ALVAC-CEA-B7.1 vaccine subcutaneously (SC) once weekly for 3 weeks.

Two weeks after the third vaccine administration, patients receive tetanus toxoid and ALVAC-CEA-B7.1 vaccine SC on day 1 and irinotecan IV over 90 minutes, leucovorin calcium IV, and fluorouracil IV on days 1, 8, 15, and 22. Treatment repeats every 6 weeks for 4 courses in the absence of disease progression or unacceptable toxicity.

* Arm II: Patients receive ALVAC-CEA-B7.1 vaccine and chemotherapy as in arm I.
* Arm III: Patients receive chemotherapy as in arm I. After completion of chemotherapy, patients with partial or complete response may receive ALVAC-CEA-B7.1 vaccine SC once weekly on weeks 1-3 and 6.

PROJECTED ACCRUAL: A total of 90 patients (30 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic colorectal adenocarcinoma
* No clinically active CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-1

Life expectancy:

* More than 6 months

Hematopoietic:

* Lymphocyte count at least 1,000/mm^3
* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* AST/ALT less than 3 times ULN (5 times ULN if liver metastases present)
* Alkaline phosphatase less than 3 times ULN (5 times ULN if liver metastases present)
* No hepatocellular dysfunction
* No cirrhosis

Renal:

* Creatinine less than 2.5 mg/dL

Cardiovascular:

* No uncontrolled coronary artery disease
* No symptomatic congestive heart failure

Pulmonary:

* No uncontrolled chronic obstructive lung disease

Gastrointestinal:

* No unsolved bowel obstruction or subobstruction
* No uncontrolled Crohn's disease
* No ulcerative colitis
* No concurrent chronic diarrhea

Immunologic:

* HIV negative
* No immunocompromised patients
* No diagnosis of altered immune function, including:

  * Lupus erythematosus
  * Sjogren's syndrome
  * Scleroderma
  * Myasthenia gravis
  * Goodpasture's disease
  * Addison's disease
  * Hashimoto's thyroiditis
  * Active Graves' disease
* No known allergy to egg products or neomycin
* No prior adverse reaction to tetanus toxoid-containing vaccines

Other:

* No significant comorbid medical function
* No uncontrolled infection
* No unstable diabetes mellitus
* No uncontrolled thyroid function abnormalities
* No other malignancy within the past 5 years except basal cell carcinoma or adequately treated carcinoma in situ of the cervix
* No other medical illness or mental status that would preclude study participation
* No prior severe toxicity to adjuvant chemotherapy
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior CEA-directed immunotherapy
* No other concurrent immunotherapy

Chemotherapy:

* At least 6 months since prior adjuvant chemotherapy
* No prior chemotherapy for metastatic disease
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent daily use of systemic steroids
* No concurrent nonsubstitutional hormonal therapy

Radiotherapy:

* No prior radiotherapy to more than 50% of all nodal groups
* No concurrent radiotherapy except for palliative purposes involving less than 20% of bone marrow reserve

Surgery:

* No prior major organ allograft
* Recovered from prior surgery

Other:

* At least 28 days since prior investigational products
* No other concurrent investigational products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-12

CONTACTS AND LOCATIONS:
Overall Officials: Howard L. Kaufman, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (13):
- United States (10):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Lombardi Cancer Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Earle A. Chiles Research Institute at Providence Portland Medical Center, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Scranton Hematology-Oncology, Scranton, Pennsylvania
- Canada (3):
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University, Montreal, Quebec

REFERENCES:
- [Result] Kaufman HL, Lenz HJ, Marshall J, Singh D, Garett C, Cripps C, Moore M, von Mehren M, Dalfen R, Heim WJ, Conry RM, Urba WJ, Benson AB 3rd, Yu M, Caterini J, Kim-Schulze S, Debenedette M, Salha D, Vogel T, Elias I, Berinstein NL. Combination chemotherapy and ALVAC-CEA/B7.1 vaccine in patients with metastatic colorectal cancer. Clin Cancer Res. 2008 Aug 1;14(15):4843-9. doi: 10.1158/1078-0432.CCR-08-0276. PMID 18676757